CLINICAL TRIAL: NCT03042910
Title: A PHASE 1, OPEN-LABEL STUDY TO ASSESS THE EFFECTS OF TALAZOPARIB ON CARDIAC REPOLARIZATION IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Assess the Effects of Talazoparib on Cardiac Repolarization in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-14; C3441005 (Other: Alias Study Number)
Record Dates: First submitted 2016-12-22; First posted 2017-02-03 (Estimated); Results first posted 2019-12-17 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Solid Tumor
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with advanced solid tumors (Experimental): Talazoparib 1 mg daily
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Talazoparib 1 mg orally once daily.
  Other Names: MDV3800; BMN673

SUMMARY:
This study is designed to evaluate the effects of talazoparib on cardiac repolarization in patients with advanced solid tumors with no available standard treatment options.

DETAILED DESCRIPTION:
For further talazoparib treatment, patients must enroll and initiate continued talazoparib treatment in a separate open label extension study within 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and willing and able to provide informed consent.
2. Histologically or cytologically confirmed advanced solid tumor with no available standard treatment options in the opinion of the investigator.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
4. Estimated life expectancy of ≥ 3 months.
5. Able to swallow the study drug, have no known intolerance to the study drug or excipients, and comply with study requirements.
6. Female patients of childbearing potential must have a negative pregnancy test at screening and must agree to use a highly effective birth control method from the time of the first dose of study drug through 45 days after last dose of study drug.
7. Male patients must use a condom when having sex with a pregnant woman or with a woman of childbearing potential from the time of the first dose of study drug through 105 days after last dose of study drug. Contraception should be considered for a nonpregnant female partner of childbearing potential.
8. Male and female patients must agree not to donate sperm or eggs, respectively, from the first dose of study drug through 105 days and 45 days after the last dose of study drug, respectively.
9. Female patients may not be breastfeeding at screening and must not breastfeed during study participation through 45 days after the last dose of study drug.

Exclusion Criteria:

1. Use of antineoplastic therapies within 21 days before day 1.
2. Use of any other investigational agent within 21 days before day 1.
3. Have not recovered (recovery is defined as National Cancer Institute Common Terminology Criteria for Adverse Events [CTCAE] grade ≤ 1) from the acute toxicities of previous therapy, except treatment related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
4. Electrolyte abnormality that has not responded to correction, including hypokalemia or hypocalcemia less than the lower limit of normal, or hyperkalemia or hypercalcemia greater than the upper limit of normal (ULN).
5. Major surgery within 14 days before day 1.
6. Diagnosis of myelodysplastic syndrome (MDS) or a hematologic malignancy.
7. Clinically significant cardiovascular disease.
8. Significant organ dysfunction.
9. Gastrointestinal disorder affecting absorption.
10. Current or anticipated use of a strong P-gp inhibitor, strong P-gp inducer, or strong inhibitor of BCRP.
11. Any condition (concurrent disease, infection, or comorbidity) that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data, in the opinion of the investigator or medical monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (18):
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - UCLA Hematology/Oncology - Burbank, Burbank, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA West Medical Pharmacy. Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - UCLA Hematology/Oncology - Pasadena, Pasadena, California
  - UCLA Hematology/Oncology - Porter Ranch, Porter Ranch, California
  - Torrance Health Association, DBA Torrance Memorial Physician Network/Cancer Care Associates, Redondo Beach, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-14

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was conducted in 4 countries from 07-Nov-2016 to 18 Dec 2017.
Groups:
- Talazoparib 1 mg QD: Talazoparib capsule was administered orally at 1 mg once daily (QD) for up to 22 days.
Period: Overall Study
Arm/Group | Talazoparib 1 mg QD
Started | 38
Treated | 37
Completed | 31
Not Completed | 7
Not completed — Adverse Event | 1
Not completed — Disease Progression | 2
Not completed — Withdrawal by Subject | 3
Not completed — Enrolled but not treated | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received any amount of talazoparib.
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: YEARS]
  Mean Age | 64.1 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 1
  Black or African American | 2
  Native Hawaiian or other Pacific Islander | 1
  Other | 2
  White | 31

OUTCOME MEASURES:

1. Primary Outcome: Time-matched Mean Change From Baseline in Corrected QT Intervals Based on the Fridericia's Correction Fomulation (QTcF)
Description: QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole.
Time Frame: Baseline (Day -1 time matched for each time point); 1, 2, 4 and 6 hours post-dose on Day 1; pre-dose on Day 2; pre-dose, 1, 2, 4 and 6 hours post-dose on Day 22
Population: Electrocardiographic analysis population: all enrolled participants who received at least 1 dose of talazoparib, and had at least 1 available baseline and 1 on-treatment electrocardiogram (ECG) data.
Measure: Mean (90% Confidence Interval); unit: millisecond (msec)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
millisecond (msec)
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | 3.9 [-0.6 to 8.4]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | 3.5 [-0.7 to 7.8]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | 1.6 [-1.3 to 4.5]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | -0.3 [-4.0 to 3.4]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | -3.5 [-8.0 to 1.1]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | -1.3 [-6.1 to 3.6]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 6.9 [2.2 to 11.5]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | 4.7 [-0.2 to 9.5]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | 3.0 [-1.4 to 7.3]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | 0.5 [-4.1 to 5.0]

2. Primary Outcome: Intercept of Predicted Linear Mixed Effects Models for Change From Baseline in QTcF Versus Plasma Talazoparib Concentrations at Day 22
Description: A linear mixed effects modeling approach was used to examine the relationship between the change from baseline in QTcF and the plasma concentration of talazoparib. The model included plasma concentration, time (categorical), and treatment with random participant effects on plasma concentration and the intercept. Equation used for modeling was: Y_lkt= μ_l+ p_t+ θ × C_lkt + W_k + D_k × C_kt + ε_lkt, where the dependent variable Y_lkt was for the l (treatment), k (participants) and t (time point). Parameter were: μ_l was the treatment specific intercept, θ was the slope, C was the concentration, W_k was the random patient effect on the intercept, D_k was the random patient effect on the slope, p_t was the time effect on the intercept and ε_lkt was the residual error.
Time Frame: Baseline (Day -1) to Day 22
Population: Pharmacokinetic-Pharmacodynamic analysis population: participants who received at least 1 dose of talazoparib, had at least 1 available baseline and 1 on-treatment ECG data, had at least 1 time-matched pair of plasma concentration and ECG measurement obtained at the same nominal time point and met the additional requirements for PK-PD analysis.
Measure: Number (95% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec | 4.6 [-3.2 to 12.5]

3. Primary Outcome: Concentration Slope of Predicted Linear Mixed Effects Models for Change From Baseline in QTcF Versus Plasma Talazoparib Concentrations at Day 22
Description: A linear mixed effects modeling approach was used to examine the relationship between the change from baseline in QTcF and the plasma concentration of talazoparib. The model included plasma concentration, time (categorical), and treatment with random participant effects on plasma concentration and the intercept. Equation used for modeling was: Y_lkt= μ_l+ p_t+ θ × C_lkt+ W_k+ D_k × C_kt+ ε_lkt, where the dependent variable Y_lkt was for the l (treatment), k (participants) and t (time point). Parameter were: μ_l was the treatment specific intercept, θ was the slope, C was the concentration, W_k was the random patient effect on the intercept, D_k was the random patient effect on the slope, p_t was the time effect on the intercept and ε_lkt was the residual error.
Time Frame: Baseline (Day -1) to Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: msec/nanogram/milliliter (msec/ng/mL)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec/nanogram/milliliter (msec/ng/mL) | -0.14 [-0.78 to 0.50]

4. Secondary Outcome: Time-matched Mean Change From Baseline in Corrected QT Intervals Based on the Bazett's Correction Fomulation (QTcB)
Description: QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | 0.6 [-3.2 to 4.4]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | 4.7 [0.4 to 9.0]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | 2.9 [-0.6 to 6.4]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | -0.4 [-4.3 to 3.5]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | -1.7 [-6.2 to 2.8]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | -2.4 [-7.0 to 2.3]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 1.1 [-3.8 to 6.0]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | 2.2 [-3.0 to 7.4]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | 1.6 [-3.3 to 6.6]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | 0.0 [-4.7 to 4.7]

5. Secondary Outcome: Time-matched Mean Change From Baseline in Heart Rate
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
beats per minute (bpm)
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | -3.0 [-6.0 to 0.1]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | 1.4 [-1.2 to 4.0]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | 1.4 [-0.8 to 3.7]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | 0.1 [-1.5 to 1.8]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | 2.3 [-0.3 to 4.9]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | -1.1 [-5.1 to 2.8]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | -6.0 [-9.3 to -2.6]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | -2.8 [-5.5 to -0.1]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | -1.4 [-4.7 to 1.8]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | -0.1 [-3.3 to 3.0]

6. Secondary Outcome: Time-matched Mean Change From Baseline in PR Interval
Description: PR interval is the time between the beginning of the P wave and the start of the QRS interval, corresponding to the end of atrial depolarization and onset of ventricular depolarization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | -2.3 [-4.3 to -0.3]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | -2.2 [-4.3 to -0.2]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | -3.2 [-5.7 to -0.7]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | -1.1 [-4.0 to 1.8]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | -4.5 [-7.1 to -1.9]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | -1.0 [-4.6 to 2.5]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 0.5 [-3.3 to 4.3]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | -0.1 [-4.0 to 3.9]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | -0.1 [-3.1 to 3.0]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | -2.4 [-5.4 to 0.6]

7. Secondary Outcome: Time-matched Mean Change From Baseline in QRS Interval
Description: QRS interval is the time from electrocardiogram Q wave to the end of the S wave, corresponding to ventricle depolarization.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | 2.9 [0.7 to 5.2]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | 2.0 [-0.6 to 4.6]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | 1.1 [-0.8 to 3.1]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | 0.9 [-1.7 to 3.6]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | 2.6 [0.3 to 4.8]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | 0.7 [-2.4 to 3.9]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 2.6 [-0.2 to 5.4]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | 1.3 [-1.8 to 4.4]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | 1.7 [-1.1 to 4.4]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | 0.7 [-2.5 to 3.9]

8. Secondary Outcome: Time-matched Mean Change From Baseline in QT Interval
Description: QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | 10.2 [1.9 to 18.4]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | 1.8 [-4.9 to 8.4]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | -0.9 [-5.4 to 3.6]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | 0.0 [-4.8 to 4.8]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | -6.5 [-13.7 to 0.8]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | 0.8 [-8.6 to 10.1]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 17.6 [9.1 to 26.0]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | 9.1 [1.4 to 16.7]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | 5.2 [-1.6 to 12.0]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | 1.2 [-6.6 to 9.0]

9. Secondary Outcome: Time-matched Mean Change From Baseline in RR Interval
Description: RR interval is the time elapsing between two consecutive R waves in the electrocardiogram.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: msec
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
msec
  Day 1, 1 hour: number analyzed (Participants) | 36
  Day 1, 1 hour | 42.9 [10.7 to 75.0]
  Day 1, 2 hours: number analyzed (Participants) | 33
  Day 1, 2 hours | -7.8 [-34.9 to 19.3]
  Day 1, 4 hours: number analyzed (Participants) | 35
  Day 1, 4 hours | -15.1 [-37.7 to 7.6]
  Day 1, 6 hours: number analyzed (Participants) | 29
  Day 1, 6 hours | 2.1 [-16.4 to 20.6]
  Day 2, pre-dose: number analyzed (Participants) | 32
  Day 2, pre-dose | -17.9 [-47.4 to 11.7]
  Day 22, pre-dose: number analyzed (Participants) | 27
  Day 22, pre-dose | 16.0 [-25.7 to 57.8]
  Day 22, 1 hour: number analyzed (Participants) | 30
  Day 22, 1 hour | 69.8 [29.3 to 110.3]
  Day 22, 2 hours: number analyzed (Participants) | 28
  Day 22, 2 hours | 30.5 [-4.3 to 65.3]
  Day 22, 4 hours: number analyzed (Participants) | 30
  Day 22, 4 hours | 15.6 [-16.2 to 47.4]
  Day 22, 6 hours: number analyzed (Participants) | 25
  Day 22, 6 hours | 4.1 [-30.9 to 39.1]

10. Secondary Outcome: Number of Participants With Treatment-emergent Abnormalities in 12-lead Electrocardiogram (ECG) Morphpology
Description: Morphological analyses were performed with regard to the ECG waveform interpretation as defined by the central ECG laboratory's cardiologist. Numbers of participants with new onsets for the following variables were counted: atrial fibrillation or flutter, second-degree heart block, third degree heart block, complete right bundle branch block, complete left bundle branch block, ST segment depression, ST segment elevation, T-wave abnormalities (negative T waves only), myocardial infarction pattern, and any new abnormal U waves. "New" was defined as "not present on any baseline ECG but present on any on-treatment ECG". Number of participants with abnormality in any of the variables were reported.
Time Frame: Baseline to Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Participants | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Findings in 12-lead Electrocardiogram (ECG) Parameters Meeting Predefined Criteria
Description: Criteria for clinically significant: Maximum QTcF >450 msec, Maximum QTcF >480 msec, Maximum QTcF >500 msec, Maximum QTcB >450 msec, Maximum QTcB >480 msec, Maximum QTcB >500 msec, Maximum QT Interval >500 msec, Maximum QTcF Increase <=30 msec, Maximum QTcF Increase 30 to <=60 msec, Maximum QTcF Increase <=60 msec, Maximum PR interval increase >200 msec and >=25%, Maximum QRS interval increase >100 msec and >=25%, Maximum heart rate increase >100 bpm and >25% and Maximum heart rate decrease <50 bpm and >25%.
Time Frame: Baseline (mean of all ECGs on Day -1 and pre-dose on Day 1) to Day 22
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Participants
  Maximum QTcF >450 msec | 5
  Maximum QTcF >480 msec | 1
  Maximum QTcF >500 msec | 0
  Maximum QTcB >450 msec | 13
  Maximum QTcB >480 msec | 2
  Maximum QTcB >500 msec | 0
  Maximum QT Interval >500 msec | 0
  Maximum QTcF increase <=30 msec | 33
  Maximum QTcF increase: 30 to <=60 msec | 4
  Maximum QTcF increase >60 msec | 0
  Maximum QTcB increase <=30 msec | 34
  Maximum QTcB increase: 30 to <=60 msec | 3
  Maximum QTcB increase >60 msec | 0
  Maximum PR interval increase >200 msec and >=25% | 0
  Maximum QRS interval increase >100 msec and >=25% | 1
  Maximum heart rate increase >100 bpm and >25% | 1
  Maximum heart rate decrease <50 bpm and >25% | 0

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Discontinuation Due to AEs, AEs of Special Interest, and Deaths
Description: An adverse event(AE)was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study drug. A serious adverse event(SAE)was an AE that resulted in: death; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect; was life-threatening (immediate risk of death); hospitalization or prolongation of existing hospitalization; or considered to be an important medical event. Treatment-emergent AEs (TEAEs) are AEs occurred on or after the administration of study drug. AEs related to study drug was any AE with at least a possible relationship to the study drug as assessed by the investigator. AEs of special interest were diagnosis of myelodysplastic syndrome (MDS) and acute myeloid leukemia (AML), and abnormal liver test results that met predefined criteria.
Time Frame: Day 1 to follow-up (30 days post last dose, i.e. up to 52 days)
Population: Safety population: all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Participants
  AEs | 28
  AEs related to study drug | 17
  SAEs | 3
  SAEs related to study drug | 1
  Discontinuations due to AEs | 0
  Deaths | 0
  AEs of special interest | 0

13. Secondary Outcome: Number of Participants With Clinically Notable Changes in Vital Signs Measurements
Description: Clinically notable changes included: High systolic blood pressure (SBP):>=155 millimeters of mercury (mmHg) with increase >=30 mmHg, low SBP <=90 mmHg with decrease >=20 mmHg, Both high and low SBP (i.e high SBP >=155 mmHg with increase >=30 mmHg and low SBP <=90 mmHg with decrease >=20 mmHg), High diastolic blood pressure (DBP):>=100 mmHg with increase >=15 mmHg), Low DBP (<=50 mmHg with decrease >=15 mmHg), Both high and low DBP, Heart rate >=100 bpm with increase >=30 bpm, Heart rate <=50 bpm with decrease >=15 bpm, Respiratory rate >=25 bpm, Respiratory rate <10 bpm, Oral body temperature >39 degree and Oral body temperature <=35 degree.
Time Frame: Screening (Day -29 to Day -2) to follow-up (30 days post last dose on Day 22)
Population: Safety population: all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Participants
  High SBP (>=155 mmHg with increase >=30 mmHg) | 0
  Low SBP (<=90 mmHg with decrease >=20 mmHg) | 2
  Both high and low SBP | 0
  High DBP (>=100 mmHg with increase >=15 mmHg) | 1
  Low DBP (<=50 mmHg with decrease >=15 mmHg) | 1
  Both high and low DBP | 0
  Heart rate >=100 bpm with increase >=30 bpm | 0
  Heart rate <=50 bpm with decrease >=15 bpm | 0
  Respiratory rate >=25 bpm | 0
  Respiratory rate <10 bpm | 0
  Oral body temperature >39 degree | 0
  Oral body temperature <=35 degree | 0

14. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory test included: hematology (hematocrit, hemoglobin, mean corpuscular volum, red blood cell count, platelet count, white blood cell count with differential [total neutrophils, eosinophils, monocytes, basophils, and lymphocytes]),chemistry (albumin, total protein, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, total bilirubin, blood urea nitrogen, creatinine, non-fasting glucose, carbon dioxide, calcium, chloride, magnesium, phosphate, potassium, sodium and lactate dehydrogenase), and additional tests (urine or serum pregnancy tests for women of childbearing potential). Clinically significant laboratory abnormality was determined by the investigator.
Time Frame: Baseline to follow-up (30 days post last dose on Day 22, i.e. up to Day 52)
Population: Safety population: all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
Participants | 3

15. Secondary Outcome: Area Under the Plasma Concentration-time Profile From Time 0 to 24 Hours After Dosing (AUC24) of Plasma Talazoparib on Day 1 and Day 22
Description: Day 22 subpopulation: amongst the participants with reported pharmacokinetic (PK) parameters on Day 22, exclusion of values from the summary statistics calculations due to dose modifications (eg, dose interruptions, dose reductions) was handled on a case by case basis, resulting in a subpopulation of participants with no prior dose modifications.
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Day 1; pre-dose, 1, 2, 4, and 6 hours post-dose on Day 22
Population: Pharmacokinetic (PK) analysis population: all participants who had sufficient concentration data to derive at least 1 PK parameter. Here, number analyzed signifies participants with available date for the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram*hour/milliliter (pg*hr/mL)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
picogram*hour/milliliter (pg*hr/mL)
  Day 1 | 54200 (42)
  Day 22: number analyzed (Participants) | 30
  Day 22 | 209000 (36)
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 208000 (37)

16. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Plasma Talazoparib on Day 1 and Day 22
Description: as for outcome 15
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Day 1; pre-dose, 1, 2, 4, and 6 hours post-dose on Day 22
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram/milliliter (pg/mL)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
picogram/milliliter (pg/mL)
  Day 1 | 4350 (47)
  Day 22: number analyzed (Participants) | 30
  Day 22 | 16300 (32)
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 16400 (32)

17. Secondary Outcome: Time for Cmax (Tmax) of Plasma Talazoparib on Day 1 and Day 22
Description: as for outcome 15
Time Frame: Pre-dose, 1, 2, 4, 6, and 24 hours post-dose on Day 1; pre-dose, 1, 2, 4, and 6 hours post-dose on Day 22
Population: Pharmacokinetic (PK) analysis population: all participants who had sufficient concentration data to derive at least 1 PK parameter.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
hour (hr)
  Day 1 | 2.00 [0.92 to 6.00]
  Day 22: number analyzed (Participants) | 30
  Day 22 | 2.00 [0.97 to 6.00]
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 2.00 [0.97 to 6.00]

18. Secondary Outcome: Predose Concentration (Ctrough) of Plasma Talazoparib on Day 22
Description: as for outcome 15
Time Frame: Pre-dose, Day 22
Population: as for outcome 17
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
pg/mL
  Day 22: number analyzed (Participants) | 30
  Day 22 | 4990 (53)
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 4950 (56)

19. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of Plasma Talazoparib on Day 22
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed. Day 22 subpopulation: amongst the participants with reported pharmacokinetic (PK) parameters on Day 22, exclusion of values from the summary statistics calculations due to dose modifications (eg, dose interruptions, dose reductions) was handled on a case by case basis, resulting in a subpopulation of participants with no prior dose modifications.
Time Frame: Pre-dose, 1, 2, 4, and 6 hours post-dose on Day 22
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour (L/hr)
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
liter/hour (L/hr)
  Day 22: number analyzed (Participants) | 30
  Day 22 | 4.8 (36)
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 4.8 (37)

20. Secondary Outcome: Accumulation Ratio (Rac) of Plasma Talazoparib on Day 22
Description: Rac was calculated as, area under the curve from time zero to end of dosing interval on Day 22 (AUCtau) divided by area under the curve from time zero to end of dosing interval on Day 1 (AUCtau). Area under the concentration curve from time 0 to end of dosing interval (AUCtau), where dosing interval was 6 hours. Day 22 subpopulation: amongst the participants with reported pharmacokinetic (PK) parameters on Day 22, exclusion of values from the summary statistics calculations due to dose modifications (eg, dose interruptions, dose reductions) was handled on a case by case basis, resulting in a subpopulation of participants with no prior dose modifications.
Time Frame: Pre-dose, 1, 2, 4, and 6 hours post-dose on Day 22
Population: as for outcome 15
Measure: Median (Full Range); unit: ratio
Arm/Group | Talazoparib 1 mg QD
Number analyzed (Participants) | 37
ratio
  Day 22: number analyzed (Participants) | 30
  Day 22 | 3.96 [1.89 to 14.4]
  Day 22 Subpopulation: number analyzed (Participants) | 27
  Day 22 Subpopulation | 3.98 [1.89 to 14.4]

ADVERSE EVENTS:
Time Frame: Day 1 to follow-up (30 days post last dose, i.e. up to 52 days)
Arm/Group | Talazoparib 1 mg QD
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 3/37
Other Adverse Events (participants affected / at risk) | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=37)
Anaemia (Blood and lymphatic system disorders) | 1
Spontaneous Haemorrhage (Blood and lymphatic system disorders) | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Syncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib 1 mg QD (N=37)
Anaemia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 9
Platelet count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT03042910/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT03042910/SAP_001.pdf